CLINICAL TRIAL: NCT05363332
Title: Impact and Sequelae of High Ventilatory Drive in Critically Ill COVID-19 Patients With Acute Respiratory Failure Requiring High Flow Oxygen or Mechanical Ventilation: Mechanistic and Genomic Characterization Using Artificial Intelligence
Brief Title: Impact and Sequelae of High Ventilatory Drive in Critically Ill COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Althaia Xarxa Assistencial Universitària de Manresa (Other); Hospital Universitario Central de Asturias (Other)
Responsible Party: Principal Investigator, Candelaria de Haro, Medical doctor and Doctor of Philosophy, Corporacion Parc Tauli
Other Study IDs: HighDrive COVID-19
Record Dates: First submitted 2022-04-29; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: COVID-19; Critical Illness; Hypoxemic Respiratory Failure; Neurocognitive Dysfunction; Mechanical Ventilation Complication
MeSH Terms: conditions — COVID-19; Critical Illness; Respiratory Insufficiency; Cognition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Cohort: Patients with a diagnosis of moderate or severe pneumonia or ARDS secondary to COVID-19.
- Non COVID-19 Cohort: Patients with a diagnosis of moderate or severe pneumonia or ARDS not secondary to COVID-19.

SUMMARY:
Critically ill COVID-19 patients with acute respiratory failure, in the intensive care unit (ICU), often feature high respiratory drive, determining large inspiratory efforts resulting in high pressures and global and regional over-distention, leading to lung injury. SARS-CoV-2 neurotropic-penetration in control centers in medulla oblongata might contribute to dysregulation and to excessively high respiratory drive observed in these patients. These pathophysiological conditions may often lead to the development of patient-ventilator asynchronies in aptients under mechanical ventilation, again leading to high tidal volumes and increased lung injury. These phenomena can contribute to prolonged duration of mechanical ventilation and ICU length of stay, but also can result in long term adverse outcomes like emotional/psychological and cognitive sequelae. All them compromising the quality of life of critically ill survivors after ICU discharge.

The investigators will conduct a multicenter study in adult critically ill COVID-19 patients with hypoxemic respiratory failure, aiming to: 1) characterize incidence and clustering of high respiratory drive by developing algorithms, 2) apply artificial intelligence in respiratory signals to identify potentially harmful patient-ventilator interactions, 3) characterize cognitive and emotional sequelae in critically ill COVID-19 survivors after ICU discharge and 4) identify sets of genes and transcriptomic signatures whose quantified expression predisposed to asynchronies and cognitive impairment in critically ill COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients with hypoxemic respiratory failure.
* Admitted to ICU.
* Mechanical ventilation or high flow nasal cannula

Exclusion Criteria:

* Neurologic patients with brainsteam affection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to ICU with acure respiratory failure secondary to COVID-19 infection and other etiologies.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Respiratory drive | From day 1 at ICU until the day were the criteria of PaFi > 300 is met, up to 30 days
  To characterize the high respiratory drive phenomena in critically ill COVID-19 patients undergoing mechanical ventilation.

SECONDARY OUTCOMES:
Cluster of high respiratory drive | From day 1 of mechanical ventilation until the day of mechanical ventilation discontinuation, up to 30 days
  To describe the incidence and clustering of high respiratory drive throughout mechanical ventilation period by the development of specific algorithms.
Artificial intelligence algorithms | From day 1 of mechanical ventilation until the day of mechanical ventilation discontinuation, up to 30 days
  To apply artificial intelligence (machine learning, deep learning, pattern/image recognition and entropy) in physiologic respiratory signals to identify potentially harmful patient-ventilator interactions.
Neurocognitive disorders | 1 month after ICU discharge and 1 year after ICU discharge
  To characterize cognitive and emotional sequelae in critically ill COVID-19 survivors at 1 month and 1 year after ICU discharge.
Gene expression | day 1 of ICU admission
  Application of massive sequencing of gene expression and circulating micro-RNA in blood samples to identify sets of genes and c-miRNA whose quantified expression is related to ventilatory asynchronies and cognitive and emotional impairment in critically ill COVID-19 patients.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Candelaria De Haro, Sabadell, Barcelona
  - Fundació Althaia, Manresa
  - Hospital Universitario Central de Asturias, Oviedo

IPD SHARING:
Plan to Share IPD: Undecided